CLINICAL TRIAL: NCT02957409
Title: PAtient RegisTry Assessing Effectiveness and Safety of HEart Failure treatmeNt With LCZ696 acrOss CaNada
Acronym: PARTHENON
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLCZ696BCA03
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Heart Failure
Keywords: Heart failure; Heart Failure with Reduced Ejection Fraction; HFrEF
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- sacubitril/valsartan: Patients diagnosed with HFrEF being treated with sacubitril/valsartan according to the Canadian product label and treatment initiation with sacubitril/valsartan within the last 3 months. The usual recommended starting dose is one tablet of 49 mg sacubitril / 51 mg valsartan taken twice daily. The target dose is one tablet of 97 mg sacubitril / 103 mg valsartan taken twice daily. Investigator/designated will document sacubitril/valsartan treatment adherence throughout the 3 years study period
  Interventions: Drug: sacubitril/valsartan

INTERVENTIONS:
Drug: sacubitril/valsartan — This study is designed as an observational, naturalistic, multicenter study in patients being treated with sacubitril/valsartan as per the Canadian product label. Treatment initiation with sacubitril/valsartan must be within the last 3 months. Sacubitril/valsartan will be used as commercially available supplies which are available as Film coated tablets in 3 dosage: 1) 24 mg sacubitril / 26 mg valsartan, 2) 49 mg sacubitril / 51 mg valsartan and 3) 97 mg sacubitril / 103 mg valsartan.
  Other Names: Entresto

SUMMARY:
The purpose of the study is to describe the heart failure with reduced ejection fraction (HFrEF) patient population receiving sacubitril/valsartan treatment.

DETAILED DESCRIPTION:
The purpose of the study is to describe the heart failure with reduced ejection fraction (HFrEF) patient population receiving sacubitril/valsartan treatment.

ELIGIBILITY:
Inclusion Criteria:

* Receiving sacubitril/valsartan as per the Canadian product label and treatment initiation within the last 3 months
* Able to communicate with investigator

Exclusion Criteria:

* Participation in a clinical trial of an investigational drug, concurrently, or within the last 30 days
* Presence of any condition that in the opinion of the investigator, prohibits patient from participating in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with HFrEF being treated with sacubitril/valsartan according to the Canadian product label. Patients are being followed/treated by Cardiologist and General Practitioners from academic institution, institution and clinic
Sampling Method: Non-Probability Sample
Enrollment: 1009 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2020-10-24 (Actual); Study Completion 2020-10-24 (Actual)

PRIMARY OUTCOMES:
Rate of all-cause hospitalization or all- cause mortality in relation to NT-proBNP or BNP levels | Up to 3 years
  The primary objective is to describe baseline NT- proBNP, or BNP levels, in relation to total all- cause hospitalization or all-cause mortality in patients with HFrEF treated with sacubitril/valsartan

SECONDARY OUTCOMES:
Percentage of patients with clinically relevant symptomatic hypotension | Up to 3 years
  Symptomatic hypotension as reported by the treating physician and defined, but not limited to, severe dizziness or fainting (syncope), lack of concentration, blurred vision, nausea, cold, clammy pale skin, and rapid shallow breathing.
Percentage of patients with clinically relevant hyperkalemia | Up to 3 years
  Hyperkalemia defined as serum potassium >5.5 mmol/L [mEq/L] after a repeated measure within one week to confirm serum potassium elevation.
Percentage of patients with clinically relevant renal impairment | Up to 3 years
  Renal impairment is defined as a decrease in eGFR of ≥40% after evaluation (verified at subsequent visit) of potentially reversible causes of renal dysfunction or end stage renal disease or need for dialysis or renal transplantation.
Percentages of patients having a BNP or NT-proBNP level | Up to 3 years
  Percentage of patients having a BNP before sacubitril/valsartan initiation will be reported; whereas, percentage of patients having NT-proBNP level at baseline and NTproBNP levels throughout the registry will be reported.
Relationship between changes in NT-proBNP and all-cause mortality | Up to 3 years
Relationship between changes in NT-proBNP and total all-cause hospitalization | Up to 3 years
Relationship between changes in NT-proBNP and renal impairment | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (30):
- Canada (30):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Maple Ridge, British Columbia
  - Novartis Investigative Site, North Vancouver, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Burlington, Ontario
  - Novartis Investigative Site, Cambridge, Ontario
  - Novartis Investigative Site, Greater Sudbury, Ontario
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, Oakville, Ontario
  - Novartis Investigative Site, Sarnia, Ontario
  - Novartis Investigative Site, Scarborough Village, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Weston, Ontario
  - Novartis Investigative Site, Chicoutimi, Quebec
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Joliette, Quebec
  - Novartis Investigative Site, Laval, Quebec
  - Novartis Investigative Site, Lévis, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Saint-Jean-sur-Richelieu, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, St-George, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec

IPD SHARING:
Plan to Share IPD: Undecided